CLINICAL TRIAL: NCT07046169
Title: Bedside Ultrasound-guided Volume Management and Discharge Timing for Patients With Heart Failure During Hospitalization: A Randomized Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pan He (Other)
Responsible Party: Sponsor-Investigator, Pan He, Associate Researcher, Yingtan City People's Hospital
Organization: Yingtan City People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: POCUS-HF study
Record Dates: First submitted 2025-06-22; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Acute Decompensated Heart Failure (ADHF)
Keywords: Heart Failure (HF); Point-of-Care Ultrasound (POCUS); Inferior Vena Cava (IVC); Pulmonary B-lines
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Active Comparator): Standard Clinical Assessment-Guided Management"
  *(Discharge based on symptoms/signs alone: Clinical congestion score ≤2 + NYHA class ≤II)
  Interventions: Other: clinical assessment
- Intervention Arm - Subgroup A (Experimental): POCUS-Guided Management (Standard Discharge Criteria) (IVC ≥1.8 mm + collapsibility >50% + B-lines ≤5, alongside clinical criteria)
  Interventions: Other: Ultrasound-Guided Volume Assessment and Decongestion Strategy (UVADS)
- Intervention Arm - Subgroup B (Experimental): POCUS-Guided Management (Strict Discharge Criteria) (IVC <1.8 mm + collapsibility >50% + B-lines ≤5, alongside clinical criteria)
  Interventions: Other: Ultrasound-Guided Volume Assessment and Decongestion Strategy (UVADS)

INTERVENTIONS:
Other: Ultrasound-Guided Volume Assessment and Decongestion Strategy (UVADS) — Unique Combination: Simultaneously tracks IVC collapsibility index (>50%) + pulmonary B-line counts (≤5) to guide therapy, unlike studies using either metric alone.Thresholds Tested: Compares ESC consensus thresholds (IVC <2.1cm) vs. exploratory Asian-optimized thresholds (IVC <1.8cm) in Subgroup B.
  Arms: Intervention Arm - Subgroup A; Intervention Arm - Subgroup B
Other: clinical assessment — Discharge based on symptoms/signs alone: Clinical congestion score ≤2 + NYHA class ≤II
  Arms: Control Arm

SUMMARY:
Brief Summary of the POCUS-HF Study

The goal of this clinical trial is to determine whether using bedside ultrasound (POCUS) to guide fluid management and discharge timing can improve outcomes for hospitalized heart failure (HF) patients. The study aims to answer the following questions:

Does POCUS-guided management (using measurements of the inferior vena cava (IVC) and lung B-lines) reduce the risk of rehospitalization and death compared to standard clinical assessment alone? What is the optimal IVC value for determining the safest discharge timing for HF patients in China and Asia?

Researchers will compare two groups:

Intervention group: Patients receive daily POCUS assessments (IVC diameter and lung B-lines) to guide fluid management and discharge decisions.

Control group: Patients receive standard care based on clinical symptoms and signs alone.

Participants will:

Undergo twice-daily POCUS measurements during hospitalization (intervention group only).

Be discharged based on either POCUS criteria (IVC and B-line thresholds) or clinical criteria (control group).

Attend follow-up visits at 7 days, 1 month, 3 months, 6 months, and 1 year after discharge to track rehospitalizations, complications, and survival.

The study hopes to provide evidence that POCUS can help reduce residual fluid overload at discharge, lower rehospitalization rates, and improve long-term outcomes for HF patients.

DETAILED DESCRIPTION:
Point-of-Care Ultrasound-Guided Volume Management During Hospitalization and Discharge Timing in Patients with Heart Failure: A Randomized Controlled Trial (POCUS-HF Study) Heart failure (HF) is a clinical syndrome caused by structural or functional abnormalities of the heart leading to inadequate perfusion of the body's organs and tissues^[1]^. It is characterized by recurrent episodes of acute decompensation requiring frequent hospitalizations and is a leading cause of hospitalization and mortality in the elderly^[2,3]^. Globally, approximately 64.34 million people are affected by HF, with about 3 million patients hospitalized annually. Approximately 25% to 30% of patients are readmitted within 30 to 90 days after discharge, and 50% are readmitted within 6 months^[4]^. The 5-year mortality rate is as high as 50%^[5]^. Recent epidemiological surveys indicate that the number of chronic HF patients in China has exceeded 8.9 million^[6]^. With an aging population and increasing chronic disease burden, the prevalence of HF continues to rise. As a significant global cause of morbidity and mortality, HF poses a major challenge to patients and healthcare systems in China, necessitating serious attention as a public health issue^[7-9]^. The high readmission rate not only increases healthcare costs and worsens prognosis but also highlights the inadequacy of current HF management strategies.

Congestion is a major reason for frequent hospitalizations in patients with acute decompensated HF and a key predictor of poor outcomes^[10,11]^, as well as an important treatment target. However, despite diuretic therapy, a significant proportion of acute HF patients still exhibit signs of congestion at discharge, which is associated with higher risks of readmission and mortality^[12,13]^. Studies show that 30-50% of acute HF patients have residual congestion at discharge, and these patients have higher rates of readmission and mortality within 1 year compared to those without congestion^[10]^. Research by Lala et al.^[14]^ similarly found that only 52% of HF patients were free of clinical congestion at discharge, yet 38% of these patients developed recurrent congestion requiring hospitalization within 60 days. Numerous clinical trials have observed that venous congestion, rather than low cardiac output, is the primary reason for HF hospitalizations^[15]^. Although current guidelines emphasize the importance of aggressive congestion management, these data suggest a lack of clear assessment strategies, leading to suboptimal volume management at discharge.

The gold standard for congestion assessment is invasive cardiac catheterization to measure right and left atrial pressures^[16]^. However, due to its invasive nature, time-consuming process, and associated risks, it is generally unsuitable for routine use in decompensated HF patients during hospitalization or pre-discharge assessment. Congestion assessment is a dynamic process involving various clinical and physiological parameters. However, guidelines do not clearly define the optimal method for assessing decongestion in HF, and current standards rely on improvements in clinical symptoms and signs as indicators of treatment efficacy and discharge readiness^[17]^. Yet, symptom and sign-based assessments can only detect moderate to severe congestion. Clinical findings such as dyspnea, orthopnea, systemic edema, elevated jugular venous pressure, and third heart sounds are important for identifying decompensated HF, but none of these signs can accurately assess the underlying hemodynamic changes causing congestion. Even patients without clinical signs of congestion may have subclinical volume overload^[4]^. Due to the dissociation between clinical manifestations and cardiac filling pressures, relying solely on clinical findings has low sensitivity and poor predictive value for identifying decompensated HF^[18]^. Therefore, for HF management, especially pre-discharge congestion assessment, combining clinical evaluation with other parameters (e.g., biomarkers, imaging) is essential to guide volume management during hospitalization and assess congestion before discharge, thereby reducing residual congestion at discharge and lowering readmission and mortality rates.

Point-of-care ultrasound (POCUS) is a non-invasive, portable, and easy-to-learn adjunct to physical examination. Inferior vena cava (IVC) imaging and lung ultrasound (LUS) can be easily performed at the bedside using portable devices. These methods provide reliable estimates of right atrial pressure and pulmonary congestion, respectively, and quickly reflect changes in volume status post-treatment. They are already widely used for fluid management in dialysis patients^[19,20]^, shock management in sepsis^[21,22]^, and HF prognosis assessment^[23-25]^. Previous studies have shown that IVC correlates well with right atrial pressure, offering high sensitivity and specificity, and outperforms physical examination in detecting elevated jugular venous pressure^[24]^. Persistently dilated IVC with low collapsibility index in HF patients at discharge predicts a higher risk of readmission. Pulmonary B-lines (ultrasound artifacts representing extravascular lung edema) correlate with the severity of pulmonary congestion. A systematic review of 13 studies found that HF patients with ≥15 B-lines at discharge had a fivefold higher risk of readmission or death^[26]^. Recently, the ESC Heart Failure Association consensus statement recommended using IVC imaging and LUS for pre-discharge assessment of residual congestion and discharge guidance. IVC diameter <2.1 mm with collapsibility >50% and fewer than 5 B-lines are proposed as key discharge criteria^[12]^. However, these recommendations are based on expert consensus and lack validation in large randomized controlled trials. A small pilot study (CAVAL US-AHF)^[4]^ demonstrated that IVC and LUS-guided HF therapy reduced subclinical congestion at discharge and improved short-term outcomes, suggesting that IVC combined with LUS is a valuable and novel approach for guiding HF treatment. However, this study had a small sample size (n=60) and focused on a Western population, where the average diuretic dose was 170 mg/day, compared to 40-60 mg/day in Chinese HF patients. Thus, the applicability of these findings to Chinese and Asian populations remains unclear. Additionally, the CAVAL US-AHF study^[4]^ used IVC and LUS only to guide decongestion therapy, not discharge timing. Further research is needed to explore the use of IVC combined with LUS for guiding discharge timing. Moreover, the IVC <2.1 mm threshold recommended by the ESC consensus is based on Western populations, and the optimal IVC value for Chinese and Asian HF patients at discharge remains unknown.

Therefore, we propose a randomized controlled trial (POCUS-HF study) to investigate the use of POCUS-assessed IVC and B-lines for guiding volume management during hospitalization in HF patients and to explore the relationship between IVC at discharge and HF risk, aiming to determine the optimal IVC threshold for discharge timing in Chinese and Asian HF patients and provide quantitative discharge criteria.

2. Research Content, Methods, and Technical Approach 2.1 Research Content

1. POCUS-guided volume management using IVC and B-line parameters during hospitalization This randomized controlled trial compares the efficacy of clinical assessment combined with POCUS (IVC and B-line metrics) versus clinical assessment alone in guiding volume management for HF patients, validating the safety and efficacy of POCUS-guided therapy.
2. Determining optimal discharge timing based on IVC Collecting IVC values at discharge to investigate their relationship with HF readmission risk and using multivariate analysis and risk prediction models to identify the optimal IVC cutoff value, providing quantitative discharge criteria for HF patients.

2.2 Key Technical Challenges

1. How to use POCUS for more precise volume management during hospitalization IVC has been shown to correlate well with right atrial pressure, offering high sensitivity and specificity, and outperforming physical examination in detecting elevated jugular venous pressure. B-lines correlate with pulmonary congestion severity. In this study, these two metrics will be measured twice daily, with diuretic doses adjusted in the intervention group to gradually reduce IVC diameter and B-line count, ensuring patients reach discharge criteria without complications like hypotension or electrolyte imbalances.
2. How to use POCUS for more precise discharge timing POCUS is a key imaging tool for volume assessment. In this study, intervention group patients will undergo POCUS assessment before discharge to evaluate volume status, providing a more precise and quantitative approach compared to clinical assessment alone. Discharge will only be permitted when volume status meets predefined criteria (IVC <2.1 mm and B-line count <5). Additionally, half of the intervention group will follow stricter discharge criteria (IVC <1.8 mm and B-line count <5) to further explore the relationship between IVC at discharge and HF prognosis.

2.3 Innovations This study addresses the clinical reality of HF patients requiring frequent readmissions due to recurrent decompensation. By combining clinical assessment with POCUS (IVC and B-line metrics), it offers a more precise and personalized approach to volume management during hospitalization and explores the relationship between IVC and readmission risk, determining the optimal discharge timing to minimize residual congestion at discharge. This provides a novel and valuable method for reducing HF readmission risk.

2.4 Technical, Economic, and Social Benefits This study aims to use POCUS to guide HF treatment and discharge timing, reducing residual congestion at discharge and lowering readmission rates, thereby improving medium- to long-term outcomes. This approach could significantly reduce patient healthcare costs and alleviate the economic burden on China's healthcare system, offering substantial socioeconomic benefits and guiding broader implementation.

2.5 Methods and Technical Approach 2.5.1 Research Methods

1. Study Design This is a prospective, single-center, single-blind, randomized, controlled trial.
2. Study Population

   A total of 150 acute decompensated HF patients (sample size calculation detailed below) will be prospectively enrolled. Key inclusion criteria:

   Hospitalized adults aged 18-90 with a diagnosis of acute decompensated HF by a cardiologist.

   Willing and able to undergo POCUS for IVC and B-line assessment. Signed informed consent and able to complete follow-up.

   Key exclusion criteria:

   Patients on invasive or non-invasive ventilation. Active lung cancer, pulmonary fibrosis, interstitial lung disease, or pneumonia.

   Chronic obstructive pulmonary disease with pulmonary hypertension or cor pulmonale.

   Cardiogenic shock. Severe renal insufficiency (creatinine clearance <30 mL/min). Severe aortic or mitral stenosis. Life expectancy <6 months. Patients undergoing ultrasound within 24 hours of admission or unable to provide consent.

   Patients discharged or transferred before meeting discharge criteria.
3. Randomization Patients will be block-randomized 1:1 to the POCUS-guided group (intervention) or clinical-guided group (control), stratified by atrial fibrillation. The intervention group will be further randomized 1:1 into subgroups A and B with different discharge criteria.
4. Blinding A single-blind design will be used, where patients are unaware of their group assignment to avoid bias. The intervention group's treatment team will be unblinded to POCUS results, while the control group's team will remain blinded.
5. Interventions All patients will undergo echocardiography within 48 hours of admission (standard HF care). Additionally, daily POCUS assessments (IVC diameter, collapsibility, and B-line count) will be performed twice daily. The intervention group's treatment will be guided by clinical and POCUS findings, while the control group will rely solely on clinical assessment.

   Discharge Criteria:

   Control group: Clinical congestion score ≤2 and NYHA class ≤II. Intervention group A: Clinical congestion score ≤2, NYHA class ≤II, IVC ≥1.8 mm with collapsibility >50%, and B-line count ≤5.

   Intervention group B: Clinical congestion score ≤2, NYHA class ≤II, IVC <1.8 mm with collapsibility >50%, and B-line count ≤5.

   POCUS Assessment:

   IVC and LUS will be performed using a Mindray ultrasound system by experienced cardiologists blinded to group assignment.
6. Follow-up Patients will be followed at 7 days, 1 month, 3 months, 6 months, and 1 year post-discharge via clinic visits or phone calls.
7. Outcomes Primary endpoint: Composite of HF readmission and cardiac death. Secondary endpoints: Acute kidney injury, hypotension, and electrolyte imbalances during hospitalization.
8. Sample Size Calculation Based on the CAVAL US-AHF study, with an expected 13% event rate in the POCUS group and 37% in the control group (α = 0.05, power = 0.80), 68 patients per group are required. Accounting for 10% dropout, 75 patients per group (total 150) will be enrolled.
9. Statistical Analysis Data will be analyzed using intention-to-treat principles. Continuous variables will be compared using t-tests or Wilcoxon tests, and categorical variables with chi-square or Fisher's exact tests. Kaplan-Meier and log-rank tests will assess event rates. Analyses will use R 4.1.2 and SPSS 28.0.
10. Quality Control To minimize bias, clinical assessors, sonographers, and outcome adjudicators will be blinded to group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis:

Hospitalized adults (age 18-90) with acute decompensated HF per ESC 2023 criteria:

Signs/symptoms (e.g., dyspnea, edema) + objective evidence (e.g., elevated NT-proBNP, imaging).

Clinical Status:

NYHA Class II-IV at admission. Systolic BP ≥90 mmHg without vasopressor support.

Technical Feasibility:

Able to undergo POCUS assessments (supine positioning, adequate acoustic windows).

Consent:

Willing to provide informed consent and complete follow-up.

Exclusion Criteria:

* Respiratory Confounders Active pneumonia, interstitial lung disease, or lung cancer (may mimic/obscure B-lines).

COPD with pulmonary hypertension (mPAP ≥25 mmHg) or cor pulmonale (alters IVC dynamics).

Cardiovascular Instability Cardiogenic shock (SBP <90 mmHg + lactate >2 mmol/L requiring inotropes). Acute coronary syndrome (STEMI/NSTEMI) within 7 days (may require alternate therapies).

Technical Barriers Subcostal scarring or abdominal dressings preventing IVC visualization. Body habitus (BMI >40 kg/m²) with persistently poor acoustic windows. Renal/Hepatic Risk AKI (KDIGO Stage 2/3) or dialysis dependence (limits diuretic responsiveness). Cirrhosis (Child-Pugh B/C) (alters volume assessment reliability). Procedural/Logistic Planned cardiac device implantation (e.g., CRT) during hospitalization. Non-adherence (inability to complete follow-up per protocol). Other Exclusions Pregnancy (physiologic IVC changes confound interpretation). Terminal illness (life expectancy <6 months unrelated to HF).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Composite rate of heart failure-related rehospitalization or cardiac death within 1 year post-discharge | Assessed at 30 days, 90 days, 6 months, and 1 year post-discharge
  Components:
  HF rehospitalization: Unplanned admission >24 hours requiring IV diuretics/vasoactive drugs.
  Cardiac death: Death from HF, MI, arrhythmia, or unexplained sudden death.

CONTACTS AND LOCATIONS:
Locations (1):
- Yingtan People's Hospital, Yingtan, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No